CLINICAL TRIAL: NCT00319254
Title: Phase II Study Of SKI-606 In Subjects With Advanced Or Metastatic Breast Cancer
Brief Title: Study Evaluating SKI-606 (Bosutinib) In Subjects With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A2-201; B1871014
Record Dates: First submitted 2006-04-24; First posted 2006-04-27 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-12

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advanced breast cancer (Experimental)
  Interventions: Drug: SKI-606 (Bosutinib)

INTERVENTIONS:
Drug: SKI-606 (Bosutinib) — SKI-606 (Bosutinib) 400mg once daily, for as long as tolerated or until disease progression.

SUMMARY:
The purpose of this study is to determine if SKI-606 (Bosutinib) is effective in the treatment of advanced or metastatic breast cancer. Patients must have current Stage IIIB, IIIC or IV breast cancer and have progressed after 1 to 3 prior chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB, IIIC or IV breast cancer not curable with available therapy.
* Patients must have progressed after 1 but not more than 3 prior chemotherapy regimens.
* Life expectancy of at least 16 weeks.
* Ability to swallow whole capsules.

Exclusion Criteria:

* Use of or requirement for bisphosphonates within 8 weeks prior to screening.
* Any other cancer within 5 years of screening, except for basal cell carcinoma or cervical carcinoma in situ
* Uncontrolled cardiac disease including congestive heart failure, angina, heart attack, etc.
* Recent or ongoing significant gastrointestinal disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (4):
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Cleveland, Ohio
- Pfizer Investigational Site, Darlinghurst, New South Wales, Australia
- France (2):
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Saint-Herblain
- Pfizer Investigational Site, Pokfulam, Hong Kong
- Pfizer Investigational Site, Floriana, Malta
- Poland (2):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Wroclaw
- Pfizer Investigational Site, Moscow, Russia
- Ukraine (3):
  - Pfizer Investigational Site, Sumy, Ukraine
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Uzhhorod

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A2-201&StudyName=Study%20Evaluating%20SKI-606%20In%20Subjects%20With%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib: Four bosutinib 100 milligram (mg) capsules, equivalent to 400 mg bosutinib orally once daily for 48 weeks, or until disease progression, unacceptable toxicity or withdrawal of consent occurred.
Period: Overall Study
Arm/Group | Bosutinib
Started | 75
Treated | 73
Completed | 21
Not Completed | 54
Not completed — Withdrawal by Subject | 4
Not completed — Death | 46
Not completed — Lost to Follow-up | 2
Not completed — Enrolled, Not Treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bosutinib
Number analyzed (Participants) | 73
Age Continuous [Mean (Standard Deviation); unit: years] | 54.27 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Rate
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from death case report forms (CRFs). Percentage of participants who had not experienced progression or death by Week 16 is reported.
Time Frame: Baseline up to Week 16
Population: Intent-To-Treat (ITT) population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 73
percentage of participants | 39.6 [28.1 to 50.8]

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) And Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 30 days after last dose of study treatment
Population: Safety population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 73
percentage of participants
  AEs | 97
  SAEs | 33

3. Secondary Outcome: Overall Survival (OS)
Description: OS was estimated by Kaplan-Meier method. Survival was defined as the time period from the date of first dose of study treatment to the date of death, censored at the participant's last contact date. Percentage of participants who were still alive at 2 years is reported.
Time Frame: Baseline up to Year 2
Population: ITT population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 73
percentage of participants | 26.4 [14.7 to 39.7]

4. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR was based on the assessment of confirmed complete remission (CR) or confirmed partial remission (PR) according to sponsor modified Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all target and non-target lesions. Confirmed PR defined as more than or equal to (>=) 30% decrease in sum of the longest dimensions (LD) of the target lesions taking as a reference the baseline sum LD. Confirmed responses are those that persist on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: Baseline up to Year 1
Population: ITT population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 73
percentage of participants | 5.5 [1.5 to 13.4]

5. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit was defined as a confirmed CR or PR, or stable disease (SD) for more than (>) 24 weeks as the best response before the first evidence of progressive disease (PD). A participant demonstrating CR, PR, or SD >24 weeks at any time while on study was counted in the numerator.
Time Frame: Baseline up to end of treatment (Week 77)
Population: ITT population included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 73
percentage of participants | 27.4 [17.6 to 39.1]

6. Secondary Outcome: Number of Participants With Change From Baseline in Laboratory Test Results
Description: Number of participants with potentially clinically significant (PCS) laboratory values are reported. Criteria for PCS laboratory values include: aspartate aminotransferase (AST), alanine aminotransferase (ALT) >5*upper limit of normal(ULN) milliunit/milliliter(mU/mL); total bilirubin >3*ULN micromole/L; sodium <130, magnesium <0.4 and >1.23 millimole/L; lipase >2*ULN microkats/L; neutrophils <1*10^9/L. Participants meeting at least 1 PCS criteria are reported.
Time Frame: Baseline up to end of treatment (Week 77)
Population: Safety population included all enrolled participants who received at least 1 dose of study treatment. Here "N" (Number of Participants Analyzed) represents number of participants who had at least 1 on-treatment assessment.
Measure: Number; unit: participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 68
participants
  Sodium (<130 mmol/L) | 2
  Magnesium (<0.4 mmol/L) | 3
  Magnesium (>1.23 mmol/L) | 3
  Total Bilirubin (>3*ULN) | 1
  ALT (>5*ULN) | 12
  AST (>5*ULN) | 10
  Lipase (>2*ULN) | 1
  Neutrophils (<1*10^9/L) | 1

7. Secondary Outcome: Number of Participants With Change From Baseline in Electrocardiogram (ECG)
Description: Number of participants with potentially clinically significant (PCS) ECG findings are reported. Criteria for PCS ECG findings include: no sinus rhythm; heart rate >=120 beats per minute (bpm) or increase >=15 bpm; QT interval corrected using Bazett's formula (QTcB) >60 milliseconds (msec) change from baseline; and overall ECG evaluation not normal.
Time Frame: Baseline up to end of treatment (Week 77)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 64
participants
  No sinus rhythm | 12
  Heart Rate (>=120 bpm and increase >=15bpm) | 2
  QTcB Interval (>60 msec change from baseline) | 1
  Overall ECG not normal | 12

8. Secondary Outcome: Number of Participants With Change From Baseline in Vital Signs, Physical Examinations, and Ophthalmological Examinations
Description: Number of participants with potentially clinically significant (PCS) vital signs and physical examinations are reported. Criteria for PCS vital signs include: respiratory rate >25 breaths/minute and PCS physical examinations include: an increase or decrease from baseline of >=7% in body weight.
Time Frame: Baseline up to end of treatment (Week 77)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Bosutinib
Number analyzed (Participants) | 54
participants
  Respiratory Rate (> 25 breaths/minute) | 6
  Weight (decrease >=7%) | 9
  Weight (increase >=7%) | 1
  Ophthalmological examinations | 0

9. Secondary Outcome: Concomitant Medications Used for Management of Adverse Events (AEs)
Description: Number of participants taking any non-study medications which were administered from Study Day 1 to last dose of study treatment (Week 77) as a management of an AE were to be reported.
Time Frame: Day 1 up to end of treatment (Week 77)
Population: Data for this pre-specified outcome measure was not statistically summarized for analysis, but collected and reported in individual participant listings as planned.
Arm/Group | Bosutinib
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Karnofsky Performance Status (KPS) at Week 1, 4, 8, 12, 16, Every 8 Weeks Thereafter and 14 Days After Last Dose of Study Treatment
Description: KPS: 11 level score ranged 100 to 0, to assess functional impairment. 100:Normal; 90:Able to carry on normal activity; 80:Normal activity with effort, some signs or symptoms of disease; 70:Cares for self, unable to carry on normal activity or to do active work; 60:Requires occasional assistance but is able to care for most of needs; 50:Requires considerable assistance and frequent medical care; 40:Disabled,requires special care and assistance; 30:Severely disabled; hospitalization indicated although death is not imminent; 20:Very sick; 10:Morbibund,fatal processes progressing rapidly; 0:Death.
Time Frame: Baseline, Weeks 1,4,8,12,16, every 8 weeks thereafter and 14 days after last dose of study treatment
Population: Data for this pre-specified outcome was collected but not statistically summarized for analysis as there were no clinically significant changes observed.
Arm/Group | Bosutinib
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Population Pharmacokinetics (PK)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Pre-dose, 2, 7, 20 hours post-dose on Day 1 of Week 4 and pre-dose on Day 1 of Weeks 1, 8, 12, 16, and 24
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bosutinib
Serious Adverse Events (participants affected / at risk) | 24/73
Other Adverse Events (participants affected / at risk) | 70/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=73)
Diarrhoea (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Oedema peripheral (General disorders) | 2
Chest discomfort (General disorders) | 1
General physical health deterioration (General disorders) | 1
Performance status decreased (General disorders) | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Coma (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib (N=73)
Anaemia (Blood and lymphatic system disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 48
Nausea (Gastrointestinal disorders) | 40
Vomiting (Gastrointestinal disorders) | 33
Abdominal pain (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 19
Asthenia (General disorders) | 14
Pyrexia (General disorders) | 7
Oedema peripheral (General disorders) | 6
Malaise (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 9
Weight decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.